CLINICAL TRIAL: NCT07143916
Title: A Satisfaction Survey for Anterior Bite Turbos in Orthodontic Patients: A Prospective Clinical Trial
Brief Title: Bonded Bite Turbos Were Bonded to Palatal Surfaces of Maxillary Incisors for Sixty Patients With Anterior Deep Overbite to Check Acceptance Rate of Patients to These Bite Turbos.
Acronym: ABT-SAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fady Hussein, professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Anterior Bite Turbos
Record Dates: First submitted 2025-07-25; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Deep Bite Malocclusion
Keywords: bite ramps; anterior bite plates; bite turbos; patient satisfaction; patient-reported outcomes
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with anterior deep overbite who needs anterior bite turbos (Experimental): Sixty patients with anterior deep bite malocclusion were treated with composite bite turbos bonded to the maxillary central incisors. A questionnaire form using the Likert scale with 5 responses (very unpleasant, unpleasant, acceptable, pleasant and very pleasant) was used by patients to document their satisfaction and feedback regarding the bite turbos after 1 week and 1 month.
  Interventions: Procedure: bonded anterior bite turbos

INTERVENTIONS:
Procedure: bonded anterior bite turbos — Sixty patients with anterior deep bite malocclusion were treated with composite bite turbos bonded to the maxillary central incisors. A questionnaire form using the Likert scale with 5 responses (very unpleasant, unpleasant, acceptable, pleasant and very pleasant) was used by patients to document their satisfaction and feedback regarding the bite turbos after 1 week and 1 month.
  Other Names: fixed bite turbos

SUMMARY:
Background: Bonded composite bite turbos are an efficient tool in the treatment of deep bite malocclusion. Patient satisfaction with orthodontic appliances has been correlated with treatment success. The aim of this study is to evaluate the level of patient satisfaction associated with bonded composite anterior bite turbos in deep bite treatment.

Materials and Methods: Sixty patients with anterior deep bite malocclusion were treated with composite bite turbos bonded to the maxillary central incisors. A questionnaire form using the Likert scale with 5 responses (very unpleasant, unpleasant, acceptable, pleasant and very pleasant) was used by patients to document their satisfaction and feedback regarding the bite turbos after 1 week and 1 month. Statistical analyses with chi-square test was used to analyze the data for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking orthodontic treatment
* Good oral hygiene
* Decreased lower anterior facial height
* Increased anterior overbite
* Full Permanent dentition
* Overjet less than 5 mm

Exclusion Criteria:

* Patients older than 25 years
* Deciduous and mixed dentition
* Patients with periodontal disease

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
assess patient satisfaction levels with anterior bite turbos | 1 week and after 1 month
  A questionnaire form using the Likert scale with 5 responses (very unpleasant, unpleasant, acceptable, pleasant and very pleasant) was used by patients to document their satisfaction and feedback regarding the bite turbos after 1 week and 1 month.
the level of patient satisfaction associated with bonded composite anterior bite turbos in orthodontic patients | patients will submit prospectively their satisfaction levels after 1 week and after 1 month after bonding the bite turbos
  A questionnaire form using the Likert scale with 5 responses (very unpleasant, unpleasant, acceptable, pleasant and very pleasant) was used by patients to document their satisfaction and feedback regarding the bite turbos after 1 week and 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Othman, A.Prof Orthodontics, Study Director — Fcaulty of Dentistry Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
is ready to share upon request

REFERENCES:
- [Derived] Fahim FH, Baumann DL, Othman A, Abdelsalam RM, Deyab HA, von See C, ElAbbasy DO. Patient Satisfaction with Anterior Bite Turbos: A Prospective Clinical Trial. Dent J (Basel). 2025 Sep 8;13(9):412. doi: 10.3390/dj13090412. PMID 41002685